CLINICAL TRIAL: NCT01901133
Title: A Phase I, Non-randomized, Open-label, Single-dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of MDV3100 in Male Subjects With Mild or Moderate Hepatic Impairment and Normal Hepatic Function
Brief Title: Hepatic Impairment Study With MDV3100 in Subjects With Mild and Moderate Hepatic Impairment Compared to a Healthy Control Group
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 9785-CL-0009
Record Dates: First submitted 2013-06-18; First posted 2013-07-17 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Pharmacokinetics of MDV3100; Healthy Subjects; Kidney Diseases
Keywords: Phase 1; MDV3100; Hepatic Impairment; Kidney Diseases; Xtandi; enzalutamide
MeSH Terms: conditions — Kidney Diseases | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Mild hepatic impairment subjects + control (Experimental)
  Interventions: Drug: MDV3100
- B: Moderate hepatic impairment subjects + control (Experimental)
  Interventions: Drug: MDV3100

INTERVENTIONS:
Drug: MDV3100 — Oral
  Other Names: Xtandi; enzalutamide

SUMMARY:
This study will assess the influence of hepatic impairment on the pharmacokinetics, safety and tolerability of a single dose of MDV3100 in male subjects.

The study will consist of two treatment arms. Arm A will assess the influence of mild hepatic impairment, and Arm B will assess the influence of moderate hepatic impairment. Data obtained from subjects with hepatic impairment will be compared to data from Body Mass Index (BMI) and age-matched subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must meet all of the following inclusion criteria:

  * Subject must be non-fertile, i.e., surgically sterilized or must practice an adequate contraceptive method to prevent pregnancies
  * Body Mass Index (BMI) of at least 18.5 and no greater than 34.0 kg/m2.
* Subjects with mild or moderate hepatic impairment must also meet the following inclusion criteria:

  * Child-Pugh classification Class A (mild, 5 or 6 points) or Class B (moderate, 7 to 9 points) liver function impairment.

Exclusion Criteria:

* All subjects must not have any of the following characteristics:

  * Known or suspected hypersensitivity to MDV3100 or any components of the formulation used.
  * History of seizure or any condition that may predispose to seizure. Also history of loss of consciousness or transient ischemic attack within 12 months of enrollment (Day 1 visit).
  * Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug (excluding non-active hay fever).
  * Abnormal pulse and/or blood pressure (BP) measurements at the pre-study visit as follows: Pulse <40 or >90 bpm; mean systolic BP >160 mmHg; mean diastolic BP >100 mmHg (BP measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured
  * A QTcF interval of >450 ms after repeated measurements (consistently after duplicate measurements), a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS).
  * Significant renal dysfunction (creatinine clearance below 60 mL/min, estimated according to the method of modification of diet in renal disease (MDRD) formula).
  * Regular use of any inducer of metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit.
  * Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half life.
* For subjects with normal hepatic function:

  * Regular use of any prescribed or OTC (over-the-counter) drugs, which includes vitamins, natural and herbal remedies (e.g. St John's wort) and food supplements in the 4 weeks prior to admission to the Clinical Unit and use of any drugs in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day).
  * Positive serology test for HBsAg, anti HAV (IgM), anti-HCV, anti-HIV-1 or anti-HIV-2.
* For subjects with mild or moderate hepatic impairment:

  * Fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period. (e.g. advanced ascites, infection of ascites, fever, active gastrointestinal bleeding).
  * Change in dose regimen of medically required medication within the last two weeks before pre-study examination (allowed co-medication in patients), and/or the use of unallowed co-medication in the 3 weeks prior to admission to the clinical unit (not allowed: any known hepatic enzyme altering agents or compounds known to restrict metabolism).
  * Presence of a hepatocellular carcinoma, or an acute liver disease caused by an infection or drug toxicity.
  * Severe portal hypertension or surgical porto-systemic shunts, including TIPSS (Transjugular intrahepatic portosystemic shunt).
  * Biliary obstruction or other cause of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
  * Signs of significant hepatic encephalopathy (Hepatic encephalopathy score >2).
  * Severe ascites and/or pleural effusion
  * Esophageal variceal bleeding in the medical history.
  * Thrombocyte level below 40x109/L and /or hemoglobin below 90 g/L.
  * Previous liver transplantation.
  * Positive serology test for, anti HAV (IgM), anti-HIV-1 or anti-HIV-2.

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetics measured by AUC0-inf following single dose of MDV3100 | Day 1 through Day 50 (25 times)
  Area under the plasma concentration - time curve extrapolated to infinity (AUC0-inf) in subjects with mild and moderate hepatic impairment to matched control subjects with normal hepatic function.
Assessment of pharmacokinetics measured by Cmax following single dose of MDV3100 | Day 1 through Day 50 (25 times)
  Maximum concentration (observed) (Cmax) in subjects with mild and moderate hepatic impairment to matched control subjects with normal hepatic function.

SECONDARY OUTCOMES:
Composite of pharmacokinetics following single dose of MDV3100 | Day 1 through Day 50 (25 times)
  Measured by Time to attain Cmax (tmax), AUC up to last quantifiable concentration (AUC0-last), Apparent terminal elimination half life (t1/2), Apparent volume of distribution during the terminal phase after extra vascular dosing (Vz/F), Apparent total body clearance after extra vascular dosing (CL/F), Cmax, t1/2, AUC0-inf, Unbound maximum concentration (observed) (Cmax,u), Unbound AUC extrapolated to infinity (AUC0-inf,u), Unbound apparent total body clearance after extra vascular dosing (CLu/F), Unbound apparent volume of distribution during the terminal phase after extra vascular dosing (Vz,u/F), Fraction unbound (fu).
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG) and clinical safety laboratory and adverse events | Day 1 through Day 50
  For hepatic impaired subjects, additional Child-Pugh classification will be performed after MDV3100 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Operation Senior Research Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Arensia, Chisinau, Moldova

REFERENCES:
- [Derived] Gibbons JA, Ouatas T, Krauwinkel W, Ohtsu Y, van der Walt JS, Beddo V, de Vries M, Mordenti J. Clinical Pharmacokinetic Studies of Enzalutamide. Clin Pharmacokinet. 2015 Oct;54(10):1043-55. doi: 10.1007/s40262-015-0271-5. PMID 25917876